CLINICAL TRIAL: NCT04370925
Title: A Multicenter Prospective Randomized Controlled Clinical Trial of Hyperthermic Intraperitoneal Chemotherapy After Colectomy in Patients With Colorectal Cancer at High Risk of Peritoneal Carcinomatosis
Brief Title: Efficacy of HIPEC in Patients With Colorectal Cancer at High Risk of Peritoneal Carcinomatosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sun Yat-sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Guangdong Provincial People's Hospital (Other); Meizhou People's Hospital (Other); First People's Hospital of Foshan (Other); Shantou Central Hospital (Other); Jiangmen Central Hospital (Other); Shenzhen Second People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); ZhuHai Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Hospital (Other Government); Peking University Cancer Hospital & Institute (Other); Peking University People's Hospital (Other); Fudan University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Chongqing University Cancer Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Wuhan University (Other); Sichuan Provincial People's Hospital (Other); West China Hospital (Other); The People's Hospital of Leshan (Other); People's Hospital of Deyang City (Unknown); Hebei Medical University Fourth Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital Of Southwest Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); The Third People's Hospital of Chengdu (Other); The Affiliated Tumor Hospital of Guangxi Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-06
Record Dates: First submitted 2020-04-08; First posted 2020-05-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Colectomy; Hyperthermic intraperitoneal chemotherapy; Peritoneal carcinomatosis
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matched control (Active Comparator): Patients undergo radical resection of primary colorectal cancer and receive standard adjuvant systemic chemotherapy
  Interventions: Procedure: Radical colectomy; Drug: Systemic chemotherapy
- HIPEC (Experimental): Patients undergo radical resection of colorectal cancer and HIPEC simultaneously or within 2 days after primary tumor resection. Followed by standard adjuvant systemic chemotherapy
  Interventions: Procedure: Radical colectomy; Procedure: HIPEC; Drug: Systemic chemotherapy

INTERVENTIONS:
Procedure: Radical colectomy — Patients undergo radical resection of the primary colorectal cancer(open or laparoscopic/robotic)
Procedure: HIPEC — HIPEC(simultaneously or within 2days after resection) with mitomycin c (30 mg/m2) at 43°C for 90 minutes.
  Arms: HIPEC
Drug: Systemic chemotherapy — Systemic chemotherapy regimens: CapeOx and mFOLFOX6 are preferred for stage Ⅲ patients.
  CapeOx:oxaliplatin 130 mg/m2 IV d1 + capecitabine 1000mg/m2 po bid d1-14. Repeat every three weeks for eight cycles.
  mFOLFOX6:oxaliplatin 85 mg/m2 IV d1 + leucovorin calcium 400 mg/m2 IV d1 + 5-FU 400 mg/m2 IV bolus d1 + 5-FU 2400 mg/m2 continuous IV over 46-48 hours d1-2. Repeat every two weeks for twelve cycles.
  For stageⅡpatiens, regimens recommend by NCCN guide line(2019 v1) are acceptable.

SUMMARY:
The purpose of this study is to determine the efficacy of adjuvant HIPEC with Mitomycin C after colectomy in the treatment of colorectal cancer patients at high risk of peritoneal carcinomatosis.

DETAILED DESCRIPTION:
The effectiveness of cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (HIPEC) have been addressed for the treatment of peritoneal carcinomatosis in selected patients. However, prophylactic HIPEC in colorectal cancer patients at high risk of metachronous peritoneal metastases remained controversial. In this study, patients with colorectal cancer cT4N0-2M0(AJCC/UICC staging system 8th edition) and planed to undergo intentionally colectomy (laparotomy, laparoscopy，or robotic ) are randomized into HIPEC group and control group. In HIPEC group, closed HIPEC is performed with Mitomycin C(30mg/m2) at 43 °C for 90 minutes, simultaneously or within 2 days after colectomy and followed by systemic chemotherapy. For the patients in the control group, systemic chemotherapy were administered after colectomy. The primary endpoint is peritoneal recurrence-free survival (pRFS) rate. Secondary end points include overall survival (OS) rate, disease free survival (DFS) rate, liver metastatic rate, toxic effects, quality of life scores. All efficacy analyses are conducted in the intention-to-treat population, per-protocol population and pT4 subgroups due to pathologic tumor invasion can not be acquired before HIPEC. Safety analysis include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Nonpregnant or breast-feeding women
* ECOG status 0-1
* Colorectal adenocarcinoma or mucinous adenocarcinoma;
* Intraoperative confirmed cT4N0-2M0 Colorectal cancer (visual determination - according to AJCC 8th edition) without previous anti-cancer treatment and R0 resection could be achieved
* Laboratory tests within 2 weeks before Randomization：Neutrophil ≥ 2.0 /mm3, , platelets ≥ 100,000/mm3, hemoglobin≥90g/l, Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ×ULN), total bilirubin(TBIL)≤ 1.5 × ULN, serum creatinine ≤ 1.5 ×ULN
* Written informed consent

Exclusion Criteria:

* Rectal cancer below peritoneal reflection
* Concurrent with or have other cancer within the past 5 years ( except for skin basal cell carcinoma, or cervical carcinoma in situ, who have received radical treatment)
* Severe abdominal infection or extensive fibrosis of peritoneal cavity that lead to impossible separation
* Surgical procedures conversion(from robotic or laparoscopic surgery to laparotomy) or emergency surgery due to perforation or obstruction
* Existence of distance metastasis during surgery (M1) or can not achieve R0 resection
* Contraindiction of mitomycin c(chickenpox or shingles)
* Poorly controlled respiratory or cardiac disease, severe hepatic or renal dysfunction,drug abuse or uncontrolled mental disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Peritoneal recurrence free survival | 3-year
  Peritoneal recurrence free survival is calculated from the date of randomization to the date of record peritoneal recurrence(with or without other metastasis), ovarian metastasis, malignant ascites, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Disease free survival | 3-year
  Disease free survival is calculated from randomization to to the date of a first relapse, the diagnosis of a secondary colorectal cancer after the initial diagnosis, or death from any cause, whichever occurred first.
Overall survival | 5-year
  Overall survival is calculated from randomization to death from any cause.
Liver metastatic rate | 3-year
  Liver metastatic rate is calculated from randomization to to the date of liver metastasis with or without other organ metastasis.
Number of participants with adverse events | Up to 1 month after the last chemotherapy cycle
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First People's Hospital of FoShan (Affiliated FoShan Hospital of Sun Yat-sen University), Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincal people's Hospital, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Six Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - JiangMen Central Hospital Affiliated JiangMen Hospital Of SUN YAT-SEN University, Jiangmen, Guangdong
  - MeiZhou People's Hospital, Meizhou, Guangdong
  - Affiliated Shantou Hospital of Sun Yat-sen University, Shantou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Zhuhai People's Hospital, Zhuhai hospital affiliated with Jinan University, Zhuhai, Guangdong
  - People's hospital of guangxi zhuang autonomous region, Nanning, Guangxi
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Union Hospital,Tongji Medical College, Huazhong Uninersity of Science and Technolgy, Wuhan, Hubei
  - Wuhan University Renmin Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Third Peoples' Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - People'S Hospital of Deyang City, Deyang, Sichuan
  - Leshan people's Hospital, Leshan, Sichuan
  - The Affiliated hospital of southwest medical university, Luzhou, Sichuan
  - The Second Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang